CLINICAL TRIAL: NCT03133377
Title: A Prospective Multicentre Phase III Randomised Controlled Trial of Early Activity and Mobilisation Compared With Standard Care in Invasively Ventilated Patients in Intensive Care
Brief Title: Treatment of Invasively Ventilated Adults With Early Activity and Mobilisation
Acronym: TEAM(III)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: National Health and Medical Research Council, Australia (Other); ANZICS Clinical Trials Group (Network); Medical Research Institute of New Zealand (Other); Intensive Care National Audit & Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TEAM U1111-1195-3567
Record Dates: First submitted 2017-04-10; First posted 2017-04-28 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Critically Ill, Mechanically Ventilated
Keywords: Early activity and mobilization, rehabilitation, intensive care
MeSH Terms: conditions — Critical Illness; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early activity and Mobilisation intervention (Experimental): Patients will be assessed daily by an ICU physiotherapist using the ICU Mobility Scale (IMS) to determine the dosage and type of active exercises the patient will receive, using the early activity and mobilisation protocol. This protocol is hierarchical, with the objective of each intervention session beginning with the highest level of activity possible for the longest time possible, which then steps down to lower levels of activity if the patient fatigues. The intervention will be administered on all days in which the patient is admitted to ICU during the index hospitalisation, censored at 28days after.
  Interventions: Behavioral: Early activity and mobilisation
- Standard of care (No Intervention): The control group will receive standard care from physiotherapy staff not involved in delivering the intervention. We have previously established that standard care in Australia for a patient receiving prolonged IMV (control group intervention) frequently involves no active exercise out of bed.

INTERVENTIONS:
Behavioral: Early activity and mobilisation — The early activity and mobilisation intervention is comprised of exercises based on a reproducible, physiological approach using both strength and functional activities
  Arms: Early activity and Mobilisation intervention

SUMMARY:
The aim of this study is to evaluate the effect of early activity and mobilisation during prolonged IMV on the composite outcome "days alive and out of hospital to day 180". The effect of the intervention on mortality, physical, cognitive and psychological function at 180 days, as well as cost-effectiveness of the intervention, will also be evaluated. The study will also explore process of care measures and baseline physiology and ICU mobility outcomes.

The hypothesis is that, in ICU patients expected to require prolonged IMV, early activity and mobilisation increases the number of days alive and at home to day 180 when compared with standard care.

DETAILED DESCRIPTION:
The TEAM Trial is a definitive phase III multi-centre randomised controlled trial in mechanically ventilated patients. Supported by compelling preliminary data, the trial will determine whether early activity and mobilisation during mechanical ventilation improves days alive and at home at 6 months compared to standard care. Recruiting 750 patients, this will be the largest trial ever conducted of early mobilisation.

Patients allocated to the early activity and mobilisation protocol (intervention group) will be assessed by a physiotherapist daily during the ICU stay to determine the highest level of mobility. This will determine the dosage and type of exercise that will be delivered, led by the physiotherapist with assistance from the multidisciplinary team. For both groups, concomitant care will be guided by the treating clinician. In addition, all post-ICU patient management will be at the discretion of the patient's ward-based treating physicians.

Patients will be randomized via web-based system and de-identified data will be collected on the following: baseline demographics; comorbidities; sedatives, analgesics, corticosteroids and neuromuscular blockers; pain/sedation/delirium scores; tracheostomy, intubation and renal replacement therapy. The intervention will be administered during the ICU stay upto 28days and the Day 180 follow up will be conducted centrally.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older.
2. Intubated and expected to remain invasively mechanically ventilated the day after tomorrow.
3. Sufficient cardiovascular stability to make mobilisation potentially possible, as indicated by:

   1. the absence of current brady-arrhythmia requiring pharmacological support
   2. a current ventricular rate ≤ 150 bpm
   3. most recent lactate ≤ 4.0 mmol/L
   4. current combined noradrenaline/adrenaline infusion rate of ≤ 0.2 mcg/kg/min, OR if noradrenaline/adrenaline infusion rate has increased by more than 25% in the last 6 hours, dose must be <0.1 mcg/kg/min.
   5. most recent cardiac index ≥ 2.0 L/min/m2 (where measured)
   6. no current requirement for VA ECMO
4. Sufficient respiratory stability to make mobilisation potentially possible, as indicated by:

   1. current FiO2 ≤ 0.6
   2. current PEEP ≤ 16 cm H20
   3. an absence of current requirement for NO, prone ventilation, neuromuscular blockers, ventilation, prostacyclin, VV ECMO or HFOV
   4. current RR ≤ 45 bpm

Exclusion Criteria:

1. Dependent for activities of daily living in the month prior to current ICU admission (gait aids are acceptable).
2. Documented cognitive impairment.
3. Proven or suspected acute primary brain pathology (e.g. traumatic brain injury, stroke, hypoxic brain injury).
4. Proven or suspected spinal cord injury or other neuromuscular disease that will result in permanent or prolonged weakness (not including ICU acquired weakness).
5. Has rest in bed orders and/or has bilateral non-weight bearing orders for the lower limbs.
6. Life expectancy less than 180 days due to a chronic or underlying medical condition.
7. Death is deemed inevitable as a result of the current illness and either the patient or treating clinical or substitute decision maker are not committed to full active treatment.
8. Unable to communicate in the official local language.
9. This is not the first ICU admission in the index hospital admission.
10. Fulfilled all inclusion criteria and none of the exclusion criteria ≥ 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Number of days alive and out of hospital | between randomisation and 180 days
  Any days spent in rehabilitation or a nursing home counted as days in hospital

SECONDARY OUTCOMES:
All-cause mortality | From date of randomisation up to180days.
Time from randomisation until death | From date of randomisation unitl date of death from all cause, censored at 180days
Ventilator-free days | From date of randomisation until day 28
  patients who die prior to day 28 will be assigned zero ventilator-free days
ICU-free days | From date of randomisation until day 28
  patients who die prior to day 28 will be assigned zero ICU-free days
Quality of life and health status measured using the European Quality of Life 5 Dimensions 5 Level (EQ5D-5L) | Assessed at 180days
Independent activities of daily living measured with Barthel Activities of Daily Living (ADL) Index and The Lawton Instrumental Activities of Daily Living Scale (IADL) | Assessed at 180days
Generic function and disability measured with the World Health Organisation's Disability Assessment Schedule (WHODAS) | Assessed at 180days

OTHER OUTCOMES:
Delirium free days | From date of randomisation until day 28
  Will be measured using CAM-ICU and RASS score
Cognitive function measured using Montreal Cognitive Assessment (MOCA-Blind) | Assessed at 180days
Psychological function measured using Hospital Anxiety and Depression scale (HADS) | Assessed at 180days
Psychological function measured using Impact of Event Scale - Revised (IES-R) | Assessed at 180 days
All-cause mortality | From date of randomisation up to 28 days
Days alive and out of hospital according to survival status | From date of randomisation up to 180 days
  Any days spent in rehabilitation or a nursing home counted as days in hospital.
Days in hospital, rehabilitation facility or nursing home according to survival status | From date of randomisation up to 180 days
  According to D180 survival status
Time from randomisation to ICU discharge | From date of randomisation up to 180 days
Time from randomisation to hospital discharge | From date of randomisation up to 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Carol Hodgson, Prof, Study Chair — ANZIC-RC
Locations (49):
- Australia (28):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St George Hospital, Sydney, New South Wales
  - John Hunter Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Mater Health, Brisbane, Queensland
  - Mater Private Hospital, Brisbane, Queensland
  - Caboolture Hospital, Caboolture, Queensland
  - The Prince Charles Hospital, Chermside West, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Rockhampton Hospital, Rockhampton, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Geelong Hospital - Barwon Health, Geelong, Victoria
  - St Vincent's Hospital Melbourne, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria
  - Cabrini Health, Melbourne, Victoria
  - Epworth Richmond, Melbourne, Victoria
  - Western Health, Melbourne, Victoria
  - Alfred Hospital, Prahran, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Fiona Stanley Hospital, Perth, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - St John of God Hospital, Subiaco, Western Australia
  - Royal Melbourne Hospital, Melbourne
- Germany (3):
  - The Charité, Berlin
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum rechts der Isar der Technischen Universität Mϋnchen, Munich
- Ireland (4):
  - Beacon Hospital, Dublin
  - St Vincent's Hospital, Dublin
  - Galway Hospital, Galway
  - Tallaght Hospital, Tallaght
- New Zealand (5):
  - Auckland City Hospital (CVICU), Auckland
  - Auckland City Hospital (DCCM), Auckland
  - Waikato Hospital, Hamilton
  - Tauranga Hospital, Tauranga
  - Wellington Hospital, Wellington
- United Kingdom (9):
  - Bristol Royal Infirmary, Bristol
  - Frimley Park Hospital, Frimley
  - University Hospital Lewisham, Lewisham
  - King's College Hospital, London
  - Nottingham University Hospitals, Nottingham
  - Royal Berkshire Hospital, Reading
  - Morriston Hospital, Swansea
  - Royal Cornwall Hospital, Truro
  - Queen Elizabeth Hospital Woolwich, Woolwich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hodgson CL, Bailey M, Bellomo R, Berney S, Buhr H, Denehy L, Gabbe B, Harrold M, Higgins A, Iwashyna TJ, Papworth R, Parke R, Patman S, Presneill J, Saxena M, Skinner E, Tipping C, Young P, Webb S; Trial of Early Activity and Mobilization Study Investigators. A Binational Multicenter Pilot Feasibility Randomized Controlled Trial of Early Goal-Directed Mobilization in the ICU. Crit Care Med. 2016 Jun;44(6):1145-52. doi: 10.1097/CCM.0000000000001643. PMID 26968024
- [Background] Tipping CJ, Harrold M, Holland A, Romero L, Nisbet T, Hodgson CL. The effects of active mobilisation and rehabilitation in ICU on mortality and function: a systematic review. Intensive Care Med. 2017 Feb;43(2):171-183. doi: 10.1007/s00134-016-4612-0. Epub 2016 Nov 18. PMID 27864615
- [Background] Iwashyna TJ, Hodgson CL. Early mobilisation in ICU is far more than just exercise. Lancet. 2016 Oct 1;388(10052):1351-1352. doi: 10.1016/S0140-6736(16)31745-7. No abstract available. PMID 27707476
- [Derived] Higgins AM, Lee YY, Bailey M, Bellomo R, Brickell K, Broadley T, Buhr H, Gabbe BJ, Gould DW, Harrold M, Hurford S, Iwashyna TJ, Serpa Neto A, Nichol AD, Presneill JJ, Schaller SJ, Sivasuthan J, Tipping CJ, Webb S, Young PJ, Hodgson CL; Treatment of Mechanically Ventilated Adults With Early Activity and Mobilization (TEAM) Study Investigators. The Cost-Effectiveness of Early Active Mobilization During Mechanical Ventilation in the ICU: An Economic Evaluation Alongside the Treatment of Mechanically Ventilated Adults With Early Activity and Mobilization (TEAM) Trial. Crit Care Med. 2025 Sep 1;53(9):e1725-e1735. doi: 10.1097/CCM.0000000000006715. Epub 2025 May 27. PMID 40439527
- [Derived] Broadley T, Serpa Neto A, Bailey M, Bellomo R, Brickell K, Buhr H, Gabbe BJ, Gould DW, Harrold M, Hurford S, Iwashyna TJ, Nichol AD, Presneill JJ, Schaller SJ, Sivasuthan J, Tipping CJ, Webb S, Young PJ, Higgins AM, Hodgson CL; TEAM Trial Investigators. Adverse events during and after early mobilisation: A post hoc analysis of the TEAM trial. Aust Crit Care. 2025 May;38(3):101156. doi: 10.1016/j.aucc.2024.101156. Epub 2025 Jan 17. PMID 39826257
- [Derived] Presneill JJ, Bellomo R, Brickell K, Buhr H, Gabbe BJ, Gould DW, Harrold M, Higgins AM, Hurford S, Iwashyna T, Neto AS, Nichol A, Schaller SJ, Sivasuthan J, Tipping C, Webb S, Young P, Hodgson CL; TEAM Study Investigators and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Protocol and statistical analysis plan for the phase 3 randomised controlled Treatment of Invasively Ventilated Adults with Early Activity and Mobilisation (TEAM III) trial. Crit Care Resusc. 2023 Oct 18;23(3):262-272. doi: 10.51893/2021.3.OA3. eCollection 2021 Sep 6. PMID 38046085
- [Derived] TEAM Study Investigators and the ANZICS Clinical Trials Group; Hodgson CL, Bailey M, Bellomo R, Brickell K, Broadley T, Buhr H, Gabbe BJ, Gould DW, Harrold M, Higgins AM, Hurford S, Iwashyna TJ, Serpa Neto A, Nichol AD, Presneill JJ, Schaller SJ, Sivasuthan J, Tipping CJ, Webb S, Young PJ. Early Active Mobilization during Mechanical Ventilation in the ICU. N Engl J Med. 2022 Nov 10;387(19):1747-1758. doi: 10.1056/NEJMoa2209083. Epub 2022 Oct 26. PMID 36286256
- See also: TEAM study website — https://www.teamtrial.org.au/